CLINICAL TRIAL: NCT06659146
Title: Prospective Study to Assess the Real-world Implementation of Thermotherapy Using wIRA (Water-filtered Infrared A Superficial Hyperthermia) in Addition to Standard of Care (SOC) Palliative Radiotherapy (RT)
Brief Title: Thermotherapy in Addition to SOC Palliative Radiotherapy
Acronym: ThermoRad wIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 327431
Record Dates: First submitted 2024-06-18; First posted 2024-10-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma; Breast Cancer Recurrent
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Head and neck squamous cell carcinoma (Experimental): 1) HNSCC i) Inoperable/incurable or recurrent/metastatic HNSCC with no previous radiotherapy treatment ii) Inoperable/incurable or recurrent/metastatic HNSCC with previous radiotherapy treatment (re-irradiation)
  Interventions: Device: Superficial hyperthermia
- Cutaneous squamous cell carcinoma (Experimental): 2) cSCC i) Inoperable/incurable or recurrent/metastatic cSCC with no previous radiotherapy treatment ii) Inoperable/incurable or recurrent/metastatic cSCC with previous radiotherapy treatment (re-irradiation)
  Interventions: Device: Superficial hyperthermia
- Locally recurrent breast cancer (Experimental): 3) LRBC locally recurrent breast cancer with previous radiotherapy treatment (re-irradiation)
  Interventions: Device: Superficial hyperthermia

INTERVENTIONS:
Device: Superficial hyperthermia — Superficial hypothermia will be delivered using a CE-marked water-filtered infrared A (wIRA) machine (hydrosun® TWH1500)

SUMMARY:
This study aims to investigate the efficacy and safety profile of superficial hyperthermia (wIRA) in addition to standard of care (SOC) palliative radiotherapy in patients with inoperable/incurable locally advanced or recurrent/metastatic HNSCC or cutaneous SCC superficial tumours not suitable for radical treatment.

The investigators will assess the best objective response rate (ORR) of patients with Inoperable/incurable or recurrent/metastatic HNSCC or cSCC with superficial lesion(s) treated with the combination of superficial hyperthermia (wIRA) and palliative radiotherapy.

DETAILED DESCRIPTION:
This study involves delivering heat treatment (thermotherapy or hyperthermia) in combination with radiotherapy (RT). Heat therapy (HT) is defined as an elevation of tissue or body temperature, and it can be used as a cancer treatment method due to the profound effect that heat has on cells. In this study, HT will be used alongside RT to enhance the effect of RT. Treatment will involve heating the tumour and the surrounding area using a specialised machine, a water-filtered infra-red-A (wIRA) superficial HT machine. HT has been shown to make cancer cells more sensitive to other cancer treatments such as RT, chemotherapy and immunotherapy and is currently in use in multiple cancer centres across Europe and Switzerland but not in the UK.

Guy's Cancer centre is the first in the UK to acquire this CE marked superficial wIRA hyperthermia machine. Our aim is to assess the real-world implementation of HT using wIRA in combination with RT in patients with cancers that are suitable for superficial hyperthermia treatment.

This is a prospective study to assess the real-world implementation of superficial hyperthermia (wIRA) in combination with SOC palliative radiotherapy in cancer patients not suitable for radical treatment and have superficial lesion(s) suitable for wIRA treatment. Three cohorts of patients will be invited:

1. HNSCC (Head and neck squamous cell carcinoma) i) Inoperable/incurable locally advanced or recurrent/metastatic HNSCC with no previous radiotherapy treatment ii) Inoperable/incurable locally advanced or recurrent/metastatic HNSCC with previous radiotherapy treatment (re-irradiation)
2. cSCC (Cutaneous squamous cell carcinoma) in the head and neck region i) Inoperable/incurable locally advanced or recurrent/metastatic cSCC with no previous radiotherapy treatment ii) Inoperable/incurable locally advanced or recurrent/metastatic cSCC with previous radiotherapy treatment (re-irradiation) LRBC
3. LRBC (locally recurrent breast cancer) with previous radiotherapy treatment (re-irradiation)

All patients consenting to the study will be treated with HT. The patients will receive hyperthermia either once a week or twice a week using hydrosun® TWH1500 with palliative radiotherapy. The patients will receive hyperthermia treatment for 1 hour before going for palliative radiotherapy as per standard of care. For patients who will undergo 20Gy/5# over one week, they will receive hyperthermia two times per week during their treatment. For patients undergoing 27Gy/6#, they will receive hyperthermia once a week for three weeks during the course of palliative radiotherapy.

Patients will be assessed during their treatment for toxicities, and rate of adverse events will be assessed by CTCAE version 5.0. Follow-ups and assessment of response will be done as per standard of care.

When appropriate, we will aim to collect biological samples from each patient for translational research (see below) including archival tumour sample, fresh tumour biopsy or resection sample when available, blood samples at different time intervals before, during and after their treatments as well as saliva and mouth swab at the same time points when appropriate. The samples will be analysed to further assess the tumour microenvironment, the peripheral immune response and to identify predictors of treatment response.

Blood samples will be collected at baseline, pre-hyperthermia treatment, post-hyperthermia treatment, 6 weeks post radiotherapy, 12 weeks post radiotherapy and at disease progression. Other samples for translational research will be collected upon the clinician's discretion and up to a total of six times. As a standard of care, patient reported outcomes are routinely collected to assess toxicity to radiotherapy treatment, and this will continue to collect for this study.

Data will be collected on the number of patients treated, adverse events experienced, outcomes on survival and disease progression, comparison with treatment not involving HT, and exploratory outcomes using biological samples.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed incurable or inoperable cancers with disease [at least one superficial lesion(s) or lymph node(s)] suitable for hydrosun® TWH1500 treatment
2. Patient undergoing standard of care palliative radiotherapy (suitable with the pre-specified dose and fractionation in the protocol
3. Aged ≥18 years old
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
5. Patient with capacity to consent

Exclusion Criteria:

1. No superficial tumour lesion or lymph node that is suitable for hydrosun® TWH1500 treatment.
2. Patients are not suitable for one of the pre-specified palliative radiotherapy dose and fractionation
3. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Real-world implementation | 24 months
  The real-world implementation of superficial hyperthermia by assessing the number of patients treated by the intervention in order to determine whether this new treatment can be implemented in a NHS cancer centre

SECONDARY OUTCOMES:
Best objective response rate | 24 months
  To assess the best objective response rate in patients receiving Thermotherapy (superficial hyperthermia) with palliative radiotherapy as part of the standard of care (SOC) by measuring the best objective response rate (ORR) (as determined by complete response rate and partial response rate according to RECIST 1.1)
Safety profile and toxicities | 24 months
  To determine the tolerability and safety profile of superficial hyperthermia in patients receiving SOC palliative radiotherapy by assessing the adverse events (CTCAE version 5.0) experienced by participants.
Median progression-free survival (PFS) and median overall survival (OS) | 24 months
  To evaluate the median progression-free survival (PFS) and median overall survival (OS) of patients. PFS= time from the start of treatment to progression or death; OS= time from the start of treatment to death.
  Patients not experiencing an event will be censored at the data last known to be alive and progression-free
Duration of objective response and locoregional control rates at 6 and 12 months | 24 months
  To assess the median duration of objective response and locoregional control rates at 6 and 12 months. The duration of response and disease control rates at 6, 12 and 24 months.
Quality of life (QoL) | 24 months
  To assess patient-reported outcome measures (PROMs) and quality of life (QoL) of patients using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30)
Efficacy between the lesion(s) treated with radiotherapy with hyperthermia with the lesion(s) treated with radiotherapy alone | 24 months
  To assess the differences in the efficacy between the lesion(s) treated with radiotherapy with hyperthermia with the lesion(s) treated with radiotherapy alone. Data to be collected by measuring the percentage of response, duration of response and disease control at 6, 12 and 24 months
Comparison of clinical outcomes with historical control | 24 months
  To compare clinical outcome of patients treated with combination of superficial hyperthermia and radiotherapy who may or may not undergo subsequent immunotherapy with the retrospective data of historical cohorts. Data will be retrospectively collected to compare outcomes from historical cohorts of similar cancer patients treated with standard of care radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kong, Principal Investigator — Clinical reader and honorary NHS consultant in clinical oncology
Locations (2):
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust, London
  - Guy's Cancer Centre, London

IPD SHARING:
Plan to Share IPD: Yes
IPDs may be shared with other researchers involved with the study and with the biobank team at Guys hospital.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available when the study begins and will be kept until the end of the study (2 years).
Access Criteria: i) Researchers directly involved with the study. ii) The biobank team appointed to the study. iii) Researchers not part of the direct care team will have access through King's Health Partners research passports, if required.

DOCUMENTS (1):
  • Study Protocol (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT06659146/Prot_000.pdf